CLINICAL TRIAL: NCT06562088
Title: A Phase I, Open-Label, Parallel, Fixed-Sequence Study to Evaluate the Effect of Repeated Administration of Rifampicin or Itraconazole on the Pharmacokinetics of HDM1002 in Healthy Adult Chinese Subjects
Brief Title: A Drug-Drug Interaction (DDI) Study of HDM1002 With Rifampicin and Itraconazole in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDM1002-105
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy Adult Subject
Keywords: HDM1002 tablet; Glucagon-Like Peptide-1 Receptor Agonists
MeSH Terms: interventions — Rifampin; Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: HDM1002 and rifampicin (Experimental): Part 1: Single dose of HDM1002
  Part 2: Once daily dose of rifampicin with single dose of HDM1002
  Interventions: Drug: HDM1002 and rifampicin
- Cohort 2: HDM1002 and itraconazole (Experimental): Part 1: Single dose of HDM1002
  Part 2: Once daily dose of itraconazole with single dose of HDM1002
  Interventions: Drug: HDM1002 and itraconazole

INTERVENTIONS:
Drug: HDM1002 and rifampicin — Administered orally
  Arms: Cohort 1: HDM1002 and rifampicin
Drug: HDM1002 and itraconazole — Administered orally
  Arms: Cohort 2: HDM1002 and itraconazole

SUMMARY:
The purpose of this study is to characterize the effect of rifampicin and itraconazole on the PK of single dose of HDM1002 in healthy adult subjects. The safety and tolerability of HDM1002 and rifampicin or itraconazole when given separately or together will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. According to the medical history, clinical laboratory test results, vital sign measurements, 12 lead ECG results, and physical examination results during the screening period, the investigator considers the subject to be in good general health.
2. Age range of 18-45 years old (including range), no limit to gender.
3. Eligible male participant weighed ≥50.0 kg, eligible female participant weighed ≥45.0 kg, and had a body mass index (BMI) within the range of 19.0 - 32.0 kg/m2 (including cut-off values).

Exclusion Criteria:

1. Participant has a history or family history of medullary thyroid cancer, thyroid C-cell hyperplasia, or multiple endocrine neoplasia type 2 (MEN2), or calcitonin≥50 ng/L during the screening period.
2. History of chronic pancreatitis or an episode of acute pancreatitis within 3 months prior to screening.
3. History of acute cholecystitis within 3 month prior to initiation of screening period.
4. Participant judged by investigator has dysphagia, diseases or conditions that affect gastric emptying, or affect the absorption of gastrointestinal nutrients, such as bariatric surgery or other gastrectomy, irritable bowel syndrome, dyspepsia, etc.
5. History of previous surgery that will affect the absorption, distribution, metabolism, and excretion of drugs or plan to undergo surgery during the study period.
6. During screening period, any abnormalities in physical examination, electrocardiogram, laboratory tests, and vital signs which are of clinically significant .
7. Taken or planned to take any drug that effect liver enzyme or transporter activity within 28 days prior to taking the investigational drug.
8. History of clinically significant cardiovascular and cerebrovascular disease within 6 months prior to screening or at the time of admission.
9. Presence of clinically significant ECG results judged by the investigator at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-16 (Estimated); Primary Completion 2024-11-19 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
AUC[0-∞] of HDM1002 | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  Pharmacokinetics (PK) parameter : Area under the curve from time 0 hour to ∞
AUC[0-24 h] of HDM1002 | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameter : Area under the curve from time 0 to 24 hour
Cmax of HDM1002 | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameter : Maximum observed concentration
AUC[0-t] of HDM1002 | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Area under the curve from time 0 to t hour
Tmax of HDM1002 | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Time to maximum plasma concentration
t1/2 of HDM1002 | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Half life
CL/F of HDM1002 | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Apparent Clearance
Vz/F of HDM1002 | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Apparent volume of distribution

SECONDARY OUTCOMES:
AUC[0-∞] of HDM1002 metabolites | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Area under the curve from time 0 hour to ∞
AUC[0-24 h] of HDM1002 metabolites | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Area under the curve from time 0 to 24 hour
Cmax of HDM1002 metabolites | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Maximum observed concentration
AUC[0-t] of HDM1002 metabolites | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Area under the curve from time 0 to t hour
Tmax of HDM1002 metabolites | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Time to maximum plasma concentration
t1/2 of HDM1002 metabolites | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters: Half life
CL/F of HDM1002 metabolites | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Apparent Clearance
Vz/F of HDM1002 metabolites | Cohort 1: Day 1-Day 5 and Day 12-Day 16; Cohort 2: Day 1-Day 5 and Day 9-Day 13
  PK parameters : Apparent volume of distribution
Adverse events (AEs) | Cohort 1: Day 1-Day 16; Cohort 2: Day 1-Day 13
  Number of subjects reporting AEs

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of anhui medical university, Hefei, Anhui, China